CLINICAL TRIAL: NCT04767009
Title: An Open-label, Multicenter, Phase II Single Arm Trial of Stereotactic Body Radiotherapy for Oligo-residual Disease After Effective Treatment With PD-1/PD-L1 Inhibitors Among Metastatic Non-small Cell Lung Cancer
Brief Title: SBRT for Oligo-residual NSCLC After Treatment With PD-1/PD-L1 Immune Checkpoint Inhibitors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-NSCLCSBRT-2
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-04

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Single Person; Drug Therapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT for oligo-residual NSCLC (Experimental)
  Interventions: Drug: PD-1/PD-L1 inhibitors (alone or in combination with chemotherapy); Radiation: SBRT

INTERVENTIONS:
Drug: PD-1/PD-L1 inhibitors (alone or in combination with chemotherapy) — Patients will receive PD-1/PD-L1 inhibitors for up to 2 years or until confirmed progression or unacceptable toxicity. PD-1/PD-L1 inhibitors will be administrated as an intravenous(IV) infusion.
Radiation: SBRT — Patients with oligo-residual NSCLC after effective treatment with PD-1/PD-L1 inhibitors will be treated with curative-intent SBRT of residual lesions. The choice of dose-fractionation regimen is at the discretion of the treating radiation oncologist. PD-1/PD-L1 inhibitors will be withheld one day before the treatment and resumed within 2 weeks after completion of SBRT.
  Other Names: Stereotactic body radiation therapy

SUMMARY:
Despite the impressive response rate to PD-1/PD-L1 immune checkpoint inhibitors, resistance inevitably develops in most patients. Stereotactic body radiation therapy (SBRT) plays a growing role in the management of oligometastatic disease. This study aims to evaluate the efficacy and safety of SBRT for oligo-residual NSCLC after effective treatment with PD-1/PD-L1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* ECOG PS 0-1.
* Patients with pathologically confirmed stage IV NSCLC by tumor biopsy and/or fine-needle aspiration.
* Negative for driver genes including EGFR, ALK, and ROS-1.
* Oligo-residual disease after effective treatment with PD-1/PD-L1 inhibitors that would be amenable to SBRT in the opinion of the investigator.
* Patients with brain metastasis are eligible if they are asymptomatic, neurologically stable, and off corticosteroids.
* Patients with a history of radiotherapy are eligible if they satisfy the following criteria:

  1. Radiotherapy administered more than 4 weeks before study entry.
  2. At least one measurable lesion outside the radiation field.
* Patients with no indications for palliative radiotherapy in the opinion of the investigator.
* Patients with a prior history of surgery are eligible if they have sufficiently recovered from the toxicity and/or complications of surgery.
* Signed informed consent for the use of fresh tumor biopsies before and during the treatment.
* Women of childbearing age and men must agree to use effective contraception during the trial.
* Life expectancy of more than 3 months.
* Adequate organ function within 1 week prior to enrollment:

  1. Adequate bone marrow function: hemoglobin ≥80g/L, white blood cell (WBC) count ≥ 4.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, and platelet count ≥ 100 * 10 ^ 9/L;
  2. Adequate hepatic function: total bilirubin < 1.5 x upper limit of normal (ULN). Note: If total bilirubin is > 1.5 x ULN, direct bilirubin must ≤ ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5 ULN;
  3. Adequate renal function: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min;
* Ability to understand and willingness to provide the informed consent.

Exclusion Criteria:

* Severe autoimmune disease: inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Wegener's granulomatosis and related vasculitides.
* Symptomatic interstitial lung disease or clinically active infectious/non-infectious pneumonitis.
* History of another malignancy or concurrent malignancy.
* Active infection, congestive heart failure, or any evidence of myocardial infarction, unstable angina pectoris or cardiac arrhythmia within 6 months prior to enrollment.
* Any evidence of severe or uncontrolled systemic diseases, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.
* Patients in whom palliative radiotherapy is indicated in the opinion of the investigator.
* Mixed small cell with non-small cell lung cancer histology.
* The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
* Patients who have received tumor vaccine; or administration of live, attenuated vaccine within 4 weeks before the start of treatment. Note: Influenza vaccination is permitted only during influenza season, while live, attenuated influenza vaccine such as FluMist is not allowed.
* Patients receiving immunosuppressive agents, or other investigational treatment. Long-term corticosteroid users are also excluded.
* Mental disorders, drug abuse, and social condition that may negatively impact compliance in the investigator's opinion.
* Prior allergic reaction or contraindications to PD-1/PD-L1 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Two years
  PFS was measured from the date of the initiation of treatment with PD-1/PD-L1 inhibitors to the date of disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death.

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | Two year
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0.
Overall Survival | Two years
  OS was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China